CLINICAL TRIAL: NCT01251458
Title: Phase I/II Study of Temsirolimus (Torisel®) as Novel Therapeutic Drug for Patients With Unresectable Hepatocellular Carcinoma (HCC)- A Correlative Study With Stathmin Over-expression
Brief Title: Hepatocellular Carcinoma (HCC)_Torisel_
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CCTU, Comprehensive Clinical Trial Unit, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC022
Record Dates: First submitted 2010-12-01; First posted 2010-12-02 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-01

CONDITIONS: Inoperable HCC
MeSH Terms: interventions — temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Torisel (Experimental)
  Interventions: Drug: Torisel

INTERVENTIONS:
Drug: Torisel — Torisel will be administered intravenously as an IV infusion over a 30-minute period in adult clinical studies.

SUMMARY:
This is a phase I/II study to evaluate dose limited toxicity and efficacy of Torisel

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed hepatocellular carcinoma that is not amenable to curative resection
* measurable disease
* Age >=18 years.
* Life expectancy of greater than 12 weeks.
* ECOG performance status <= 2
* Prior systemic therapy for HCC is allowed
* Adequate haematologic, renal and hepatic function
* Absence of cirrhosis or Child's A cirrhosis
* Fasting total cholesterol <9.1 mmol/liter and fasting triglyceride level <4.5 mmol/liter)

Exclusion Criteria:

* Patients who have had systemic therapy or radiotherapy within 3 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 3 weeks earlier.
* Patients receiving any other investigational agents concurrently.
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Uncontrolled intercurrent diseases such as, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
• To establish the maximum tolerated dose (MTD) and a suitable dose for Phase II evaluation of Torisel® given as a weekly dose in patients with advanced hepatocellular carcinoma (HCC) | 2 years

SECONDARY OUTCOMES:
• To determine and establish the safety and toxicity profile of Torisel® and to identify any dose limiting toxicities (DLTs) in advanced HCC | 2 Years
• To determine progression-free survival (PFS) in patients with advanced hepatocellular carcinoma (HCC) treated with Torisel® | 4 Years
• To correlate stathmin expression in pre-treatment HCC tumour biopsies and clinical response to Torisel® | 2 years
• To determine the response rate (CR and PR) based on RECIST criteria | 2 years
• To determine clinical benefit rate (CBR, percent of patients experiencing CR, PR or SD ≥ 12 weeks) | 2 years
• To determine duration of response (DR) | 2 years
• To determine overall survival (OS) | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Winnie Yeo, MD, FRCP, Principal Investigator — Department of Clinical Oncology, The Chinese University of Hong Kong
Locations (1):
- Department of Clinical Oncology, Prince of Wales Hospital, Hong Kong, Hong Kong